CLINICAL TRIAL: NCT02409381
Title: Clinical Trial, Multicenter, Phase IV, Open, Randomized, Parallel, Controlled, Non-inferiority, to Evaluate the Efficacy and Safety of Motore® Compared to Alivium® in the Treatment of Adults With Knee Osteoarthritis
Brief Title: Extract of Curcuma Longa Complexed With Phosphatidilcholine(Motore®)in the Treatment of Adults With Knee Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ache Laboratorios Farmaceuticos S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACH-MTR-04(02/13)
Record Dates: First submitted 2015-04-01; First posted 2015-04-06 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-06

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motore (Experimental): Curcuma longa complexed with phosphatidylcholine - 250 mg (Motore®), two (02) capsules orally every twelve (12) hours
  Interventions: Drug: Motore
- Alivium (Active Comparator): Ibuprofen 600 mg (Alivium®), one (01) coated tablet orally, every six (06) hours.
  Interventions: Drug: Alivium

INTERVENTIONS:
Drug: Motore — 250 mg
  Other Names: Group 1
  Arms: Motore
Drug: Alivium — 600 mg
  Other Names: Group 2
  Arms: Alivium

SUMMARY:
Prospective, multicenter, phase IV, open, randomized, parallel, controlled, in which 288 (two hundred and eighty-eight) participants of both sexes, aged between 40 and 75 years will be randomly allocated to one of two treatment groups , and treatment group 01 will be the dried extract of Curcuma longa complexed with phosphatidylcholine (Motore®), and treatment group 02 will ibuprofen (Alivium®).

DETAILED DESCRIPTION:
This study evaluate the efficacy and safety of Dry Extract of Curcuma Longa complexed with phosphatidilcholine (Motore®) Compared to Ibuprofen (Alivium® ) in the treatment of adults with knee osteoarthritis. The study population will consist in participants of both sexes, aged between 40 and 80 years old with a clinical diagnosis of knee osteoarthritis (tibiofemoral joint) based on clinical and radiological criteria (Grades 2 and 3 Kellgren and Lawrence) and who had osteoarthritis symptoms in the last six (06) months preceding the start of the study. They will be randomly allocated to one of two treatment groups , and treatment group 01 will be the dried extract of Curcuma longa complexed with phosphatidylcholine (Motore®), and treatment group 02 will ibuprofen (Alivium®).

ELIGIBILITY:
Inclusion Criteria:

* Participants of both sexes;
* Age greater than or equal to 40 years and less than or equal to 75 years;
* Clinical diagnosis of osteoarthritis of the knee (tibiofemoral joint) based on clinical and radiological criteria (Grade 2 and 3 Kellgren and Lawrence) as specified below:
* Pain on movement in the affected knee on most days of the last month, with at least partial relief at rest;
* Presence of osteophytes of at least 1 mm in radiological imaging, a report issued by a qualified professional from the center;
* Symptoms of osteoarthritis in the last 06 months preceding the start of the study;
* Visual Analogue Scale with 40mm or greater value (considering the data obtained at the randomization visit);
* Ability to understand and consent to participate in this clinical study, manifested by signing the Informed Consent Form (ICF).

Exclusion Criteria:

* Any finding of clinical observation (clinical and physical examination) or laboratory finding that is interpreted by the researcher as a medical risk to participation in the clinical trial;
* Any finding of ECG examination the investigator physician considers risk as to the research participant about their participation in the clinical trial;
* Known hypersensitivity to the components of the medications used during the study;
* Women in pregnancy or nursing period;
* in premenopausal women who do not agree to use acceptable contraceptive methods (oral contraceptives, injectable contraceptives, hormonal implants, barrier methods, abstinence, hormonal patch and tubal ligation); except surgically sterile (bilateral oophorectomy or hysterectomy);
* concomitant arthropathy that may confuse or interfere with pain assessment or efficacy, including: inflammatory arthropathy (rheumatoid arthritis, systemic lupus erythematosus, spondyloarthropathy, psoriatic arthritis, polymyalgia rheumatic), gouty arthritis, acute episodes of monoarthritis compatible with pseudogout, Paget's disease with involvement of the joint study, history of septic arthritis, avascular necrosis or intra-articular joint studied, Wilson's disease, hemochromatosis, alkaptonuria, primary osteochondromatosis fracture;
* Infectious Arthritis as gonococcal and syphilitic;
* History of significant collateral ligament injury, or anterior cruciate, or the meniscus of the joint study, requiring surgery or immobilization for more than three weeks (minor ligament injuries, six months prior to the study, are not exclusion criteria );
* History of arthroscopy of the affected knee during the six months preceding the entry of the research participant in the study;
* History of any illness that, in the opinion of the investigator, might confound the results of the study or research participant put on additional risk;
* Treatment with corticosteroids as follows:
* Use of corticosteroids orally or intramuscularly for one month prior to the randomization visit (V0);
* Administration of intra-articular corticosteroid, the joint study in the previous three months at randomization visit (V0);
* Administration of intra-articular corticosteroids in any joint a visit prior to randomization (V0) month;
* intra-articular injection of hyaluronic acid in the joint or congeners studied in the last twelve months prior to randomization visit (V0);
* Implementation of any other medical treatment for osteoarthritis in the pre-randomization visit (V0) months;
* Body Mass Index (BMI) equal to or greater than 35;
* Participant that is in use Prohibited Drug;
* the presence of serious psychiatric illness of any kind that prevents the proper performance of study-related procedures and good adherence to treatment;
* Participant that has some relation to the second degree of kinship or relationship with employees or employees of Sponsor and Research Center.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2015-06; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Reduction in the pain domain score of the WOMAC questionnaire | After 42 (forty two) days of treatment
  The primary efficacy endpoint will be the reduction in the pain domain score of the WOMAC questionnaire after 42 (forty two) days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Rocha, MD, Principal Investigator — Artroclinica de Fortaleza
Locations (1):
- Ache Laboratorios Farmaceuticos, Guarulhos, São Paulo, Brazil